CLINICAL TRIAL: NCT01550653
Title: Liraglutide Effects on Memory in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Dr. med. Volker Ott, Principal Investigator, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Ott-NN-001
Record Dates: First submitted 2012-03-01; First posted 2012-03-12 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Memory; GLP-1; Liraglutide; energy output; Memory facilitation; GLP-1 analogue
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): See "Intervention"
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator): See "Intervention"
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: liraglutide — Subcutaneous self-administration of liraglutide(Victoza)by pen. The starting dose is 0.6 mg once daily(day 0 to 7), followed by 1.2 mg once daily (day 8 to 35).
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study examines the hypothesis, that subcutaneous administration of liraglutide, an analogue of the incretin glucagon-like peptide 1, over 5 weeks improves memory functions in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-35 years
* Body mass index between 19 and 25 kg/m2
* Non-smoker

Exclusion Criteria:

* Receipt of any drug within 4 weeks prior to this trial
* Any known acute or chronic disease of the brain, heart, lung, kidney,liver, pancreas or gastrointestinal tract, any metabolic, endocrine or psychiatric disease.
* Brady- and Tachycardia, i.e. heart rate < 50 and > 90 beats per minute.
* Hypertension (systolic blood pressure > 150 mmHg, diastolic blood pressure > 90 mmHg).
* Hyperlipidemia (cholesterol, LDL, triglyceride > two times the upper reference limit based on analysis from the central laboratory)
* Impaired hepatic function measured as alanine aminotransferase (ALAT) > two times the upper reference limit based on analysis from the central laboratory
* Impaired renal function measured as creatinine > 120 µmol/l based on analysis from the central laboratory
* Family history of diabetes
* History of any eating disorder
* Known or suspected allergy to trial products
* History of drug or alcohol abuse within the last five years prior to screening

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the immediate and delayed recall of a declarative memory task (word list recall) at time points indicated in "time frame" section. | Day -7 (immediate Recall 1), Day 0 (Delayed Recall 1), Day 1 (Immediate Recall 2), Day 7 (Delayed Recall 2), Day 28 (Immediate Recall 3), Day 35 (Delayed Recall 3)
Change from baseline in the immediate and delayed recall of an Episodic Memory Task (story recall) at the time points indicated in the "Time Frame" - section. | Day -7 (immediate Recall 1), Day 0 (Delayed Recall 1), Day 28 (Immediate Recall 2), Day 35 (Delayed Recall 2)
Change from baseline in performance on a two-dimensional object location task on day 1 and day 35. | Day -7, Day 1, Day 35
Change from baseline in performance on a working-memory task on day 1 and day 35. | Day -7, Day 1, Day 35
  Digit Span Test
Change from baseline in immediate and delayed recall of a procedural memory task at the time points indicated in the "Time Frame" - section. | Day -7 (immediate Recall 1), Day 0 (Delayed Recall 1), Day 28 (Immediate Recall 2), Day 35 (Delayed Recall 2)
  Finger tapping test

SECONDARY OUTCOMES:
Change from baseline in resting metabolic rate on day 7, 28 and 35. | Day 0 , Day 7 , Day 28 , Day 35
  indirect calorimetry
Change from baseline in serum/plasma concentrations of parameters involved in glucose metabolism on day 1,7,28, and 35. | Day -7, 1, 7, 28, 35

CONTACTS AND LOCATIONS:
Overall Officials: Volker Ott, MD, Principal Investigator — University of Luebeck, Department of Neuroendocrinology
Locations (1):
- University of Luebeck, Department of Neuroendocrinology, Lübeck, Germany